CLINICAL TRIAL: NCT01580917
Title: Dynamic Plantar Microvascular Skin Response to Compressive Loads in At-risk Diabetic and Healthy Control
Brief Title: Dynamic Plantar Microvascular Skin Response to Compressive Loads in At-risk Diabetic and Healthy Control: a Pilot Study
Acronym: ILH
Status: Completed | Type: Observational
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Other Study IDs: TUSPM-JF-01
Record Dates: First submitted 2012-04-17; First posted 2012-04-19 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Foot Ulcer, Diabetic
Keywords: laser doppler anemometry; dynamic testing of tissue mechanical property; diabetic foot complications; ulcer genesis
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Diabetic Test: Diabetic individuals with a history of previous plantar ulcer and a high risk of developing a foot ulceration
- Healthy Controls: Non-diabetic, healthy individuals with low risk of developing a neurogenic foot ulcer

SUMMARY:
The purpose of this pilot study is to compare the dynamic response of microcirculation in the skin on the bottom of the big toe after applying controlled plantar stress in 25 diabetic subjects with a history of foot ulcer and 25 age-matched healthy controls to better understand the role of local hypoxia in neuropathic foot ulceration in subjects with diabetes.

The investigators hypothesize that if they apply a gait simulating load to the plantar foot and measure microvascular function, diabetic individuals will demonstrate an increased delay in reestablishing microvascular flow compared to healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* between ages 40 and 75
* history of diabetic neuropathic plantar ulcer (test subjects)
* no history of diabetes (control subjects)
* no peripheral sensory neuropathy (control subjects)

Exclusion Criteria:

* amputation or surgery on right Great Toe

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A community sample
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2007-11; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Latency time after occlusive loading | approximately 2.75 minutes after start of collection protocol
  The time between removal of occluding pressure and the initiation of the post-occlusive hyperemic response as measured by laser Doppler.

SECONDARY OUTCOMES:
Response time to baseline | 2.75 seconds after start of collection protocol
  The time interval between the start of post-occlusive hyperemic response and when the response curve reaches the baseline, or reference, flow level as measured by laser doppler.
Response time to Maximum Flow | At least 2.75 seconds after the start of collection protocol.
  The time interval between the start of the post-occlusive hyperemic response and the time to reach maximum flow as measured by laser doppler

CONTACTS AND LOCATIONS:
Overall Officials: Jinsup Song, DPM, PhD, Study Director — Temple University; James A Furmato, DPM, PhD, Principal Investigator — Temple University
Locations (1):
- Temple University School of Podiatric Medicine Gait Study Center, Philadelphia, Pennsylvania, United States